CLINICAL TRIAL: NCT02931643
Title: Postprandial Effects of Mixed Herbs and Spices on Pathways Associated With Glucose Homeostasis and Inflammation on PBMCs of Healthy Subjects - Molecular Insights Through Integration of Transcriptomics of Peripheral Blood Mononuclear Cells (PBMC) and Circulating miRNA
Brief Title: Postprandial Effects of Mixed Herbs and Spices on Pathways Associated With Glucose Homeostasis and Inflammation on PBMCs of Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Anti-Diabetic Food Centre (Other)
Responsible Party: Principal Investigator, Yoghatama Cindya Zanzer, MSc, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LUND-AFCSTAGE4-SPICEMULTIOMICS
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Spices; Functional food; Cardiometabolic risk; Metabolic syndrome; Inflammation; Peripheral blood mononuclear cell; Acute; miRNA
MeSH Terms: conditions — Metabolic Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fat challenge breakfast (Placebo Comparator): High fat breakfast without mixed-spices (% Energy Carbohydrate:Fat:Prot / 20:60:20), acute study / one time administration
  Interventions: Other: High fat challenge breakfast
- High fat challenge breakfast with mixed-spices (Experimental): High fat breakfast with mixed-spices (% Energy Carbohydrate:Fat:Prot / 20:60:20), acute study / one time administration
  Interventions: Other: High fat challenge breakfast with mixed-spices

INTERVENTIONS:
Other: High fat challenge breakfast — In this intervention, subjects are asked to consume high fat breakfast without mixed-spices. Standardized high fat breakfast corresponding to % Energy of Carbohydrate:Fat:Prot / 20:60:20
  Arms: High fat challenge breakfast
Other: High fat challenge breakfast with mixed-spices — In this intervention, subjects are asked to consume high fat breakfast with mixed-spices. Standardized high fat breakfast corresponding to % Energy of Carbohydrate:Fat:Prot / 20:60:20
  Arms: High fat challenge breakfast with mixed-spices

SUMMARY:
This study aims to investigate the effect of mixed of herbs and spices on gene expression of pathways associated with glucose homeostasis, oxidative stress, inflammation and its interrelation with circulating miRNA, in the postprandial phase in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* BMI 23-33 kg/m2
* Must be able to accept spices
* Agreed and signed informed consent

Exclusion Criteria:

* Below 18 years old
* Uncomfortable speaking English and/or difficulties in understanding spoken English
* Smoking or using snuss
* Vegetarian or vegan
* Having food allergies
* Stressed by venous blood sampling or previous experience of being difficult to be cannulated
* Receiving any drug treatment that may influence the study outcomes
* Pregnancy or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (0 hr) in untargeted PBMC gene expression profile at 4 hr | Prior to the initial intervention at 0 hr and after intervention at 4 hr
  The venous blood samples will be taken for isolation of peripheral blood mononuclear cells. Extracted total RNA will then be used for running RNA-microarray (Illumina, San Diego, CA, USA)

SECONDARY OUTCOMES:
Postprandial appetite ratings after acute intervention | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 and 240 min.
  Appetite will be assessed using standard subjective 100 mm VAS (visual analogue scale) at respective time frame throughout each visit. Appetite questionnaire includes following questions: How hungry do you feel?, How strong is your desire to eat?, How satiated (i.e. pleasantly satisfied) are you?, How full do you feel?, How much food do you think you can (or would want to) eat?, How thirsty are you?
Postprandial gastrointestinal tolerance ratings after acute intervention | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 and 240 min.
  Gastrointestinal tolerance will be assessed using standard subjective 100 mm VAS (visual analogue scale) at respective time frame throughout each visit. Gastrointestinal tolerance questionnaire includes following questions: Do you experience any abdominal pain?, Do you experience any rumbling noises in your stomach?, Do you experience any flatulence (generation of excessive gas)?, Do you experience any bloated (swollen) feeling in the abdomen?, Do you experience any acid reflux (heartburn)?, Do you experience nausea?, Do you experience an urge to vomit?
Postprandial blood glucose after acute intervention | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 and 240 min.
  The capillary blood samples will be taken for blood glucose analysis.
Postprandial insulin after acute intervention | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 and 240 min.
  The venous blood samples will be taken for insulin analysis. Insulin analysis will be conducted with routine hospital analysis at Labmedicine Skåne.
Postprandial triacylglycerol after acute intervention | Prior to the initial intervention at 0 min and after intervention at 30, 60, 90, 120, 180 and 240 min.
  The venous blood samples will be taken for plasma triacylglycerol analysis. Plasma triacylglycerol analysis will be conducted with routine hospital analysis at Labmedicine Skåne.
Postprandial non-esterified fatty acids (NEFA) after acute intervention | Prior to the initial intervention at 0 min and after intervention at 30, 60, 90, 120, 180 and 240 min.
  The venous blood samples will be taken for serum NEFA analysis. Serum NEFA analysis will be conducted with routine hospital analysis at Labmedicine Skåne.
Postprandial total cholesterol after acute intervention | Prior to the initial intervention at 0 min and after intervention at 30, 60, 90, 120, 180 and 240 min.
  The venous blood samples will be taken for plasma total cholesterol analysis. Plasma total cholesterol analysis will be conducted with routine hospital analysis at Labmedicine Skåne.
Postprandial high density lipoprotein (HDL)-cholesterol after acute intervention | Prior to the initial intervention at 0 min and after intervention at 30, 60, 90, 120, 180 and 240 min.
  The venous blood samples will be taken for plasma HDL-cholesterol analysis. Plasma HDL-cholesterol analysis will be conducted with routine hospital analysis at Labmedicine Skåne.
Postprandial low density lipoprotein (LDL)-cholesterol after acute intervention | Prior to the initial intervention at 0 min and after intervention at 30, 60, 90, 120, 180 and 240 min.
  The venous blood samples will be taken for plasma LDL-cholesterol analysis. Plasma LDL-cholesterol analysis will be conducted with routine hospital analysis at Labmedicine Skåne.
Postprandial interleukin (IL)-6 after acute intervention | Prior to the initial intervention at 0 min and after intervention at 120 and 240 min.
  The venous blood samples will be taken for serum interleukin IL-6 analysis. Serum IL-6 analysis will be conducted with routine hospital analysis at Labmedicine Skåne.
Postprandial interleukin (IL)-10 after acute intervention | Prior to the initial intervention at 0 min and after intervention at 120 and 240 min.
  The venous blood samples will be taken for serum interleukin IL-10 analysis. Serum IL-10 analysis will be conducted with routine hospital analysis at Labmedicine Skåne.
Postprandial tumor necrosis factor (TNF)-alpha after acute intervention | Prior to the initial intervention at 0 min and after intervention at 120 and 240 min.
  The venous blood samples will be taken for serum TNF-alpha analysis. Serum TNF-alpha analysis will be conducted with routine hospital analysis at Labmedicine Skåne.
Postprandial lipid peroxidation (MDA equivalent) after acute intervention | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 and 240 min.
  The venous blood samples will be taken for lipid peroxidation (MDA) assay.
Postprandial total antioxidant capacity after acute intervention | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 and 240 min.
  The venous blood samples will be taken for total antioxidant capacity (FRAP) assay.
Change from Baseline (0 hr) in untargeted circulating miRNA profile at 4 hr | Prior to the initial intervention at 0 hr and after intervention at 4 hr
  The venous blood samples will be taken for isolation of peripheral blood mononuclear cells. Extracted total RNA will then be used for running miRNA (Affymetrix, Santa Clara, CA, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Yoghatama Cindya Zanzer, MSc PhDcand, Principal Investigator — Lund University; Elin Östman, PhD A/Prof, Principal Investigator — Lund University; Congyu Xue, BSc, Study Chair — Lund University
Locations (1):
- Food for Health Science Centre, Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Antidiabetic Food Centre - VINNOVA Excellence Centre in Research and Innovation at Lund University, SWEDEN — http://portal.research.lu.se/portal/sv/projects/antidiabetic-food-centre(3a9bae87-b64a-49f5-97a4-868a8bb776ae).html